CLINICAL TRIAL: NCT05279066
Title: A Clinical Validation Study for Measuring Cardiac Output and Ejection Fraction Using a Wrist-worn Device.
Brief Title: Validation of Ejection Fraction and Cardiac Output Using Biostrap Wristband
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Ali Nsair, MD, Associate Clinical Professor, University of California, Los Angeles
Other Study IDs: 21-001030
Record Dates: First submitted 2022-01-27; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure
Keywords: ejection fraction; cardiac output
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients scheduled to undergo an elective cardiac ultrasound: All cardiac patients undergoing an elective cardiac ultrasound as an outpatient at UCLA may be asked to participate in the study. The investigators will identify eligible patients from their medical record. If interested, patients will be consented prior to their scheduled ultrasound.
  Interventions: Device: Biostrap Wristband
- Patients with a pulmonary arterial catheterization scheduled or completed: All patients hospitalized in the cardiac ICU at UCLA with a pulmonary arterial catheterization scheduled or completed may be asked to participate in the study. The investigators will identify eligible patients from their medical record. If interested, patients will be consented during their hospital stay.
  Interventions: Device: Biostrap Wristband

INTERVENTIONS:
Device: Biostrap Wristband — The Biostrap Wristband device is a non-invasive optical sensor that monitors changes in arterial pulse volume using Photoplethysmography (PPG). PPG is frequently used in wearable sensors to detect heart rate as well as other metrics such as heart rate variability (HRV) and respiratory rate. The raw biosignals recorded by the wristband device will be further processed to estimate the ejection fraction and cardiac output.

SUMMARY:
In this study, the investigators will compare the accuracy of the Biostrap wristband, a wearable device with a clinical-grade Photoplethysmography (PPG) sensor, to measure ejection fraction and cardiac output in patients undergoing a cardiac ultrasound and pulmonary arterial catheterization, respectively.

DETAILED DESCRIPTION:
This in an introductory clinical study with both cardiac patients undergoing elective cardiac ultrasound and cardiac ICU patients with pulmonary arterial catheters featuring Biostrap wristband. This is a single site, non-blinded, non-randomized study. The wristband is a wearable device that contains a clinical-grade Photoplethysmography (PPG) sensor which will measure parameters quasi-continuously and non-invasively. The device, Biostrap wristband, will measure cardiac ejection fraction (EF) and cardiac output (CO). We will enroll a total of 100 patients: 2 groups of 50. 50 patients undergoing an elective cardiac ultrasound as part of their routine medical care will wear the device for 1-2 hours as an outpatient depending on the duration of the test. 50 hospitalized patients with a scheduled or completed pulmonary arterial catheter inserted as part of their standard medical care will wear the device for 7 days.

The investigators will perform a retrospective analysis comparing the accuracy of EF and CO measured by the device in comparison to those from a 'reference device', which is the cardiac ultrasound for ejection fraction and the pulmonary arterial catheter for cardiac output values. Cardiac Ultrasound and pulmonary arterial catheters are standard of care procedures.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age.
2. Subjects who are undergoing elective cardiac ultrasound as an outpatient for group 1 or are scheduled for/completed a pilmonary arterial catheterization for group 2.
3. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Subject is unable or unwilling to wear the wristband for the required duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and woman over the age of 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Association between obtained PPG waveforms and recorded ejection (EF) fractions | 6 months
  Patients scheduled to undergo a cardiac ultrasound will wear the Biostrap wristband for the duration of the echocardiogram (1-2 hours) and a PPG waveform will be obtained from the device. The ejection fraction (measured in units of %) will also be obtained from the echocardiogram report. Then, the Artificial Intelligence (AI) staff member will do a predictive model to try and estimate the EF based on the PPG waveform. PPG-derived outcome measures will be derived from a two-step process of raw data collection followed by application of waveform derivative algorithms. They will perform an in-depth beat shape analysis of the PPG waveform that includes identifying dozens of features and critical points of each beat to derive the Ejection fraction (calculated in units of %).
Association between obtained PPG waveforms and recorded cardiac outputs (CO) | 6 months
  Patients scheduled to undergo a pulmonary arterial catheterization in the cardiac ICU will wear the biostrap wristband for 7 days and a PPG waveform will be obtained from the device. The cardiac output values (measured in units of mL and recorded using the PA catheter) will also be obtained from the patient's medical record. Then, the Artificial Intelligence (AI) staff member will do a predictive model to try and estimate the CO based on the PPG waveform. PPG-derived outcome measures will be derived from a two-step process of raw data collection followed by application of waveform derivative algorithms. They will perform an in-depth beat shape analysis of the PPG waveform that includes identifying dozens of features and critical points of each beat to derive the Cardiac Output (calculated in unites of mL).

CONTACTS AND LOCATIONS:
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States